CLINICAL TRIAL: NCT06189066
Title: Long COVID Ultrasound Trial [LOCUS Trial]
Brief Title: Long COVID Ultrasound Trial
Acronym: LOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SecondWave Systems Inc. (Industry)
Collaborators: University of Minnesota (Other); MCDC (United States Department of Defense) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00020251; W911QY-21-9-0036 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2023-12-31; First posted 2024-01-03 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Long Covid
Keywords: long covid; covid-19; long-haul COVID; post-COVID conditions (PCC); post-acute COVID-19; post-acute sequelae of SARS-CoV-2 infection (PASC); ultrasound; ultrasound stimulation; ultrasound treatment; ultrasound therapy
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Ultrasound Group (Experimental)
  Interventions: Device: Splenic Ultrasound

INTERVENTIONS:
Device: Splenic Ultrasound — Daily ultrasound application to the spleen of approximately 18 minutes per day, 5 days per week for up to 8 weeks, in addition to standard clinical care.
  Other Names: SecondWave Systems investigational MINI device

SUMMARY:
The research objective is to assess the safety and potential efficacy of spleen ultrasound stimulation as an intervention for Long COVID in a pilot study.

Specific Aims include:

* Measure Long COVID disease activity before, during and after an 8-week course of spleen-directed daily ultrasound stimulation.
* Measure molecular correlates of Long COVID disease activity before, during and after an 8-week course of spleen-directed daily ultrasound stimulation.
* Track adverse events throughout the study to assess safety of the ultrasound intervention.

DETAILED DESCRIPTION:
Ultrasound is widely used in human medicine because it is safe, non-invasive, and painless. The same kind of ultrasound that is used for imaging (for example, to visualize babies in utero) may be able to treat inflammatory diseases including Long COVID.

In Long COVID, there can be a state of hyperinflammation that persists in those with symptoms months to years after infection. This hyperinflammatory state includes elevated proinflammatory cytokines such as interferon β (IFN-β), IFN-λ1, IFN-γ, CXCL9, CXCL10, interleukin-6 (IL-6), IL-8, IL-1β , and Tumor Necrosis Factor (TNF-α) in those with Long COVID. Prolonged inflammation in those with Long COVID plays a key role in its pathogenesis and in driving the persistent symptoms.

This study will employ investigational ultrasound devices produced by SecondWave Systems called the MINI ultrasound system.

This is a pilot single-arm intervention study in which up to 15 study participants will receive noninvasive splenic ultrasound therapy over eight weeks (five daily stimulation sessions per week). Participants will be enrolled in the study for a total of 12 weeks starting at Week 0. They will undergo a 4-week Baseline Period during which no intervention is delivered to determine how study outcomes may change over time. Then, after baseline outcomes are measured at Week 4, the investigational ultrasound interventional period will begin. Outcomes will be compared from baseline at Week 4 through the end of the 8-week intervention period at Week 12. Investigational splenic-ultrasound therapy will be delivered with the SecondWave MINI ultrasound system. The objective of the study is to assess the safety and potential efficacy of spleen ultrasound stimulation as an intervention for Long COVID in a pilot study.

For ultrasound stimulation, a small wearable ultrasound device is positioned on the upper left abdomen area over the ribs. Study personnel will use an ultrasound imaging device to locate the spleen and to position the wearable MINI device in a proper location around the ribs area. Daily stimulation consists of an approximately 18-minute period for application of ultrasound to the spleen. Collection of long-COVID outcome data, patient-reported assessments, and blood draws collected at the 6 study visits to assess biomarkers of inflammation will be performed in each participant throughout the study. Stool samples will be collected at 4 timepoints to assess changes in microbiome and metabolomics over the study period. Movement activity and sleep monitoring will be collected throughout the day and correlated with other study outcomes.

The study's primary outcome measure is the endurance shuttle walk test (ESWT) and the secondary outcome measure is the Chalder fatigue scale (CFQ-11). We will also investigate exploratory outcomes that will include other activity outcomes (e.g., total movement per day, sleep patterns), vital signs (e.g. heart rate and blood pressure), biomarker assessments (e.g., CRP, ESR, cortisol), cytokine assessments, microbiome and metabolomic related assessments, and device usability and experience assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years at the time of enrollment
2. Prior diagnosis of COVID-19 by report, PCR, or home kit
3. Symptoms present for 12 or more weeks that are independent prior to SARS-CoV-2 infection including fatigue and one or more of:

   1. Myalgia or general aches/pains
   2. Joint pain
   3. Dizziness/lightheadedness
   4. Cognitive dysfunction (brain fog)

Exclusion Criteria:

1. Candidate who is unable or unwilling to postpone taking new medications used for treating Long COVID during the study period
2. Candidate that is currently taking immune modifying medications and unable to maintain stable levels of their immune medication regimen throughout the study period
3. History of intubation secondary to COVID-19
4. ICU admission for COVID-19
5. Pre-existing Lung conditions such as chronic obstructive pulmonary disease (COPD), interstitial lung disease (ILD), or severe asthma
6. Pregnant
7. History of coronary artery disease (CAD)
8. History of stroke
9. History of severe anemia of hemoglobin less than 8 g/dl
10. Prior history of Lyme disease
11. Prior history cognitive impairment
12. Any non-marijuana drug abuse history within 30 days
13. Current use of an investigational drug
14. History of prior myalgic encephalomyelitis or chronic fatigue syndrome (ME/CFS)
15. History of alcohol abuse: greater than 2 drinks a day for men and 1 drink for females
16. Prior history of postural orthostatic tachycardia syndrome (POTS)
17. Chronic fatigue secondary to any condition other than COVID-19.
18. Fibromyalgia
19. History of prior chronic pain
20. History of chronic liver disease such as cirrhosis
21. History of splenic pathology such as spleen infarct/splenomegaly
22. History of splenectomy
23. History of Sickle disease with splenic pathology
24. Taking non-approved treatments for Long COVID
25. Participant does not speak English
26. Participant is an active member of the military (service member) or DoD personnel (including civilian employees)
27. Any other clinical reasons deemed by the investigators of the study in which the patient would not be an appropriate candidate for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Within-arm change in the endurance shuttle walk test (ESWT) from baseline to the completion of an up-to 8-week intervention period. | 8 weeks
  ESWT is a standardized, externally controlled, constant-paced walking test for the assessment of endurance capacity. Improvement in this outcome will be determined by an increase of distance walked and/or increase in time walked before failure to maintain the controlled walking pace.

SECONDARY OUTCOMES:
Within-arm change in the Chalder fatigue scale (CFQ-11; Likert score) from baseline to the completion of an up-to 8-week intervention period. | 8 weeks
  CFQ-11 is a is a self-administered questionnaire for measuring the extent and severity of fatigue.
Track adverse events throughout the study to assess the safety of the ultrasound intervention. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Farha Ikramuddin, M.D., Principal Investigator — University of Minnesota Medical School, Department of Rehabilitation Medicine
Locations (1):
- University of Minnesota - Phillips-Wangensteen Building, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goggins E, Inoue H, Okusa MD. Neuroimmune Control of Inflammation in Acute Kidney Injury and Multiorgan Dysfunction. J Am Soc Nephrol. 2025 Dec 1;36(12):2473-2484. doi: 10.1681/ASN.0000000813. Epub 2025 Jul 7. PMID 40622772